CLINICAL TRIAL: NCT01217671
Title: A Phase II/III, Double-Blind, Randomized, Placebo-Controlled, Multicenter, International Study Evaluating the Safety and Efficacy of Inhaled, Human, Alpha-1 Antitrypsin (AAT) in Alpha-1 Antitrypsin Deficient Patients With Emphysema
Brief Title: International Study Evaluating the Safety and Efficacy of Inhaled, Human, Alpha-1 Antitrypsin (AAT) in Alpha-1 Antitrypsin Deficient Patients With Emphysema
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kamada, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Kamada-AAT (inhaled) 007
Record Dates: First submitted 2010-09-15; First posted 2010-10-08 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2016-04

CONDITIONS: Emphysema
Keywords: Pulmonary, Emphysema; Alpha-1 Antitrypsin Deficiency
MeSH Terms: conditions — Emphysema; alpha 1-Antitrypsin Deficiency | interventions — Inhalation; alpha 1-Antitrypsin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alpha-1 Antitrypsin (Experimental)
  Interventions: Biological: Kamada AAT for inhalation
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Kamada AAT for inhalation — Alpha-1 Antitrypsin (AAT)
  Other Names: Alpha-1 Proteinase Inhibitor (API)
  Arms: Alpha-1 Antitrypsin
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomised , placebo controlled, double blind , multicentre, Phase II/III study evaluating the safety and efficacy of Kamada AAT for inhalation in patients with Emphysema caused by Alpha-1 Antitrypsin (AAT) deficiency.

DETAILED DESCRIPTION:
Alpha-1 Antitrypsin Deficiency, also called Alpha-1-Proteinase Inhibitor (API) deficiency, is a genetic disorder characterized by the production of an abnormal amount of AAT protein and reduced circulating levels of this protein. Subjects with AAT deficiency are at increased risk for developing Emphysema. It is believed that this is the result of the chronic activity of elastase released by cells continually present in the lungs in low numbers.

Three blinded interim analyses have shown that there are no safety issues and no concerns regarding tolerability.

ELIGIBILITY:
Principal Inclusion Criteria:

* Diagnosis of emphysema confirmed by CT scan. If a report of past CT scan is not available at site documenting then a CT scan is to be performed at screening
* Male or female patients at least 18 years of age.
* Able and willing to sign an informed consent.
* Patient with record of congenital AAT deficiency of phenotype PiZZ (homozygote) or other rare phenotypes related to AAT deficiency and with AAT serum level ≤ 11 micromole. For patients receiving IV AAT augmentation therapy the serum AAT level threshold does not apply.
* FEV1/SVC <70% of predicted value post bronchodilator (SVC is slow VC) and FEV1 < 80% of predicted value post-bronchodilator
* History of at least two moderate or severe exacerbations that required change in treatment (antibiotics, systemic steroids, hospitalization) in the last 18 months prior to date of screening , with at least one of these occurring within the last 12 months prior to screening.
* Ability to comply with completion of electronic diary.
* Ability to self-administer inhaled AAT.
* No significant abnormalities in serum hematology, serum chemistry and serum inflammatory / immunogenic markers according to the Principal Investigator's judgment, taking into considerations the potential effects of the AAT deficiency.
* No significant abnormalities in urinalysis according to the Principal Investigator's judgment, taking into considerations the potential effects of the AAT deficiency.
* No significant abnormalities in ECG per investigator judgment.
* Negative for HBsAg and for antibodies to HCV, HIV-1.
* AAT deficient patients who are either naïve (not receiving IV augmentation therapy) or AAT deficient patients (receiving IV augmentation therapy), if they have been stable on regular therapy for at least 3 months prior to the screening visit and are willing to continue the same regime throughout this trial. Note that only sites in Germany can recruit patients who are currently being treated with IV AAT.Patients who stopped IV augmentation treatment 6 months prior to screening date and will not re-start this treatment for the course of the study will be considered Naïve.
* Non-pregnant, non-lactating female patients, whose screening pregnancy test is negative and who are using contraceptive methods deemed reliable by the investigator, or who are at least 2 years post-menopausal or surgically sterilized.

Principal Exclusion Criteria:

* FEV1 >= 80% or FEV1 < 20% of predicted value post-bronchodilator.
* FEV1/SVC>=70%
* History of lung transplant.
* Any lung surgery within the past two years.
* On any thoracic surgery waiting list.
* End of last exacerbation less than 6 weeks prior to screening/re-screening visit.
* Clinically significant intercurrent illnesses (except for respiratory or liver disease secondary to AAT deficiency), including: cardiac, hepatic, renal, endocrine, neurological, hematological, neoplastic, immunological, skeletal or other) that in the opinion of the investigator, could interfere with the safety, compliance or other aspects of this study. Patients with well-controlled, chronic diseases could possibly be included after consultation with the treating physician and the sponsor.
* Active smoking during the last 12 months from screening date.
* Pregnancy or lactation.
* Woman of child-bearing potential not taking adequate contraception deemed reliable by the investigator.
* Presence of psychiatric/ mental disorder or any other medical disorder which might impair the patient's ability to give informed consent or to comply with the requirements of the study protocol.
* Evidence of ongoing viral infection with HCV, HBV and/or HIV.
* Evidence of alcohol abuse or history of alcohol abuse or illegal and/or legally prescribed drugs.
* IgA Deficiency
* History of life threatening allergy, anaphylactic reaction, or systemic response to human plasma derived products.
* Participation in another clinical trial within 30 days prior to baseline visit.
* Inability to attend scheduled clinic visits and/or comply with the study protocol.
* Any other factor that, in the opinion of the investigator, would prevent the patient from complying with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2009-12; Primary Completion 2014-11 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Exacerbation events and lung density | Approximately 1 year

SECONDARY OUTCOMES:
Adverse Events | Approximately 1 year
Vital Signs | Approximately 1 year
Physical Examination | Approximately 1 year
ECG | Approximately 1 year
Lung function | Approximately 1 year
Laboratory Evaluations | Approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jan Stolk, Professor, Principal Investigator — LUMC, Leiden, Netherlands
Locations (12):
- Canada (2):
  - Inspiration Research Limited, Toronto
  - Seymour Health Centre, Vancouver
- Gentofte Hospital, Hellerup, Denmark
- Germany (2):
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Universitatsklinikum Gieben und Marburg, Marburg
- Beaumont Hospital, Dublin, Ireland
- LUMC, Leiden, Netherlands
- Sweden (2):
  - Malmo University Hospital, Malmo
  - Karolinska Universitetssjukhuset Solna, Stockholm
- United Kingdom (3):
  - Queen Elizabeth Hospital, Birmingham
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Brompton Hospital, London

REFERENCES:
- [Result] Stolk J, Tov N, Chapman KR, Fernandez P, MacNee W, Hopkinson NS, Piitulainen E, Seersholm N, Vogelmeier CF, Bals R, McElvaney G, Stockley RA. Efficacy and safety of inhaled alpha1-antitrypsin in patients with severe alpha1-antitrypsin deficiency and frequent exacerbations of COPD. Eur Respir J. 2019 Nov 21;54(5):1900673. doi: 10.1183/13993003.00673-2019. Print 2019 Nov. PMID 31467115
- See also: PubMed — https://www.ncbi.nlm.nih.gov/pubmed/31467115